CLINICAL TRIAL: NCT06502067
Title: Efficacy of Serratus Posterior Superior Intercostal Plane Block (SPSIPB) on Perioperative Analgesia and Inflamatory Markers in Breast Surgery
Brief Title: Efficacy of Serratus Posterior Intercostal Plane Block for Analgesia and Inflammatory Marker in Breast Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD94/2024
Record Dates: First submitted 2024-07-06; First posted 2024-07-15 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Breastcancer; Perioperative Pain; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- will receive serratus posterior superior block using bupivacaine (Active Comparator): between the SPSM and the 3rd rib after using a test dose of 1- 2 mL saline and Following hydro-dissection,30ml 0.25%bupivacaine will be injected.
  Interventions: Drug: Analgesia mangement group A,B
- Arm B: (control group) patients will only receive general anesthesia without block. (Other): Narcotic postoperative
  Interventions: Drug: Analgesia mangement group A,B

INTERVENTIONS:
Drug: Analgesia mangement group A,B — 1gm of paracetamol, 30mg of ketorolac and 1mg Granitryl will be given twenty minutes before the end of the operation .

SUMMARY:
To study the efficiacy of serratus posterior superior block in controlling perioperative breast cancer surgery pain and its effect on inflamatory markers.

DETAILED DESCRIPTION:
Back ground The presence of pain during the initial course of treatment in women with early-stage breast cancer was associated with significantly higher levels of c-reactive protein(CRP) ,interleukin-7(IL-7)and interleukin-13(IL-13) There is evidence of effectiveness of regional block in controlling inflamatory markers Serratus posterior superior intercostal plane block (SPSIPB) is a novel Regional technique that provides analgesia in the hemithorax, shoulder, and back of the neck which proved its efficacy in controlling pain after Video assisted thoracoscopic surgery there are little epidemiological data on (SPSIPB)usage in masectomy and lumpectomy procedures and its effect on inflamatory markers

Methodology:

* Type of the Study: Randomized prospective comparative controlled double-blinded study

  * Study Setting: Ain Shams University Hospitals
  * Study Period: One year after approval of the protocol.
  * Place :Ain shams university hospitals
  * Study Population: Adult patients who will undergo breast cancer surgey.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing unilateral breast surgery under general anesthesia
* Age 21 to 60 years with body mass index (BMI)=18 to 25 kg/m2
* American Society of Anesthesiologists (ASA) grade I-III.

Exclusion Criteria:

* Patients with Long-time use of analgesic drugs
* Past history of chest surgery,
* Allergy to local anesthetics,
* Systemic infection,
* Cognitive and language disorders precluding participation,
* Patients with coagulopathy,anticoagulant users
* hemodynamic unstable patients
* Patients with neurology, spinal, psychiatry diseases
* infection at block site
* patients refused to participate in the study .

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
is to calculate total perioperative analgesia consumption throughout (24hours). | 24 hour postoperative